CLINICAL TRIAL: NCT04198636
Title: A Randomized, Double-blind, Single-dose, Parallel-group Study to Compare the Pharmacokinetics, Pharmacodynamics, Safety and Immunogenicity of LY01011 and Xgeva® in Healthy Adults
Brief Title: A Study to Evaluate LY01011 and Xgeva® in Healthy Adults
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Luye Pharma Group Ltd. (Industry)
Collaborators: Shang Dong Boan Biotechnology Co., Ltd (Co-sponsor) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LY01011/CT-CHN-102
Record Dates: First submitted 2019-12-07; First posted 2019-12-13 (Actual); Last update posted 2019-12-13 (Actual); Status verified 2019-12

CONDITIONS: Healthy Adults
Keywords: Compare; Pharmacokinetics; Pharmacodynamics; Safety; Immunogenicity; LY01011; Xgeva®; Healthy adults
MeSH Terms: interventions — Denosumab; Injections

STUDY DESIGN:
Intervention Model Description: Parallel assignment
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LY01011 (Experimental): LY01011 injection (120mg) by subcutaneous injection once on the first day subcutaneous injection of 120 mg (1.7 ml)only once
  Interventions: Drug: LY01011
- Xgeva® (Active Comparator): Xgeva® injection (120mg) by subcutaneous injection once on the first day subcutaneous injection of 120 mg (1.7 ml)only once
  Interventions: Drug: Xgeva 120 MG in 1.7 ML Injection

INTERVENTIONS:
Drug: LY01011 — LY01011 injection (120mg) by subcutaneous injection once on the first day subcutaneous injection of 120 mg (1.7 ml)only once
  Other Names: subcutaneous injection of 120 mg (1.7 ml)
  Arms: LY01011
Drug: Xgeva 120 MG in 1.7 ML Injection — Xgeva® injection (120mg) by subcutaneous injection once on the first day subcutaneous injection of 120 mg (1.7 ml)only once
  Other Names: subcutaneous injection of 120 mg (1.7 ml)
  Arms: Xgeva®

SUMMARY:
A randomized, double-blind, single-dose, parallel-group study to compare the pharmacokinetics, pharmacodynamics, safety and immunogenicity of LY01011 and Xgeva® in healthy adults

DETAILED DESCRIPTION:
This is a phase I, randomized, double-blind, single-dose, parallel-group clinical trial .

The primary objective is to assess the pharmacokinetic similarity of single and subcutaneous injections of LY01011 or Xgeva® in healthy volunteers.

The secondary objective are to compare the safety, tolerability, immunogenicity and pharmacodynamics of single and subcutaneous injections of LY01011 or Xgeva® in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Sign the informed consent form and fully understand the test content, process and possible adverse reactions, and be able to complete the study according to the test plan requirements
2. During the study period, the subjects and partners agreed to use reliable contraceptive measures
3. Aged ≥18 years or ≤50 years, male or female (including the boundary value)
4. Male body weight≥50kg，female body weight≥45kg，and 18.0≤BMI≤28.0 kg/m2
5. Clinical laboratory examination, chest X-ray, abdominal B-ultrasound, electrocardiogram, physical examination, vital signs and various examinations are normal or abnormal without clinical significance at screening

Exclusion Criteria:

1. Subjects are suffering from or have had osteomyelitis or osteonecrosis of the Jaw, or plan to have invasive dental or maxillofacial surgery during the study, or dental or oral surgery wounds unhealed
2. Have fractures in past six months
3. The medicines that may affect bone turnover are used before screening or planned to use in the study period , including but not limited : Denosumab, bisphosphonates or fluorides were used in past 12 months; Contraceptives with hormone were used in past 6 months，Hormone replacement therapy（tibolone、hormone、selective estrogen receptor modulators）Aromatase inhibitors, calcitonin, strontium salt, parathyroid hormone (or derivative), vitamin D supplement，Anabolic steroids, systemic glucocorticoids, calcitriol or analogues, diuretics, anticonvulsant drugs；Inhalation or local use of glucocorticoids within 2 weeks
4. Hypocalcemia or hypercalcemia，or serum calcium calibrated by serum albumin was not within the normal range
5. Subjects with allergic constitution (allergic to more than two drugs or food) or known to be allergic to the ingredients of the investigational product
6. Donated whole blood, blood component, or massive hemorrhage （>450ml）three months before screening
7. Use of any vaccines in 4 weeks of initiation of study therapy
8. Use Rx or OTC drugs or nutritional health products or herbal supplements within 14 days before the screening
9. Have been playing strenuous sports in 2 weeks before screening; or other factors affecting drug absorption, distribution, metabolism, excretion
10. The average daily smoking amount is more than 5 cigarettes per day during three months before screening;
11. History of drug abuse or alcohol abuse (drank more than 14 units / week of alcohol: 1 unit =285ml beer, 25ml spirits or 100ml Wine)；
12. History of drug abuse within 5 years prior to screening, or urine drug screening test was positive；
13. other clinically significant diseases (such as neuropsychiatric system, cardiovascular system, urinary system, digestive system, respiratory system, metabolic endocrine system, blood system, skin diseases, immune diseases, tumors, etc.)
14. Any of HBsAg, HCV-Ab, Anti-HIV, TP-Ab was positive
15. Acute disease or combination of medication from the screening to the study before the use of investigational product ,
16. Take any alcoholic product within 48 hours before using the investigational product
17. Participation in another clinical trial within 3 months prior to enrollment
18. Anticipated of partner pregnancy during the study.
19. Other conditions that the investigator thinks unsuitable in this study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 168 (Estimated)
Dates: Start 2019-12-16 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Cmax | 168 days
  Assess the Cmax similarity of single and subcutaneous injections of LY01011 or Xgeva® in healthy volunteers
AUC0-t | 168 days
  Assess the AUC0-t similarity of single and subcutaneous injections of LY01011 or Xgeva® in healthy volunteers

SECONDARY OUTCOMES:
AE | 168 days
  Number of patients with treatment related adverse events assessed by change from baseline
ADA | 168 days
  Number of patients with ADA
Nab | 168 days
  Number of patients with Nab
AUC0-∞ | 168 days
  Assess area under the Curve (AUC)
Tmax | 168 days
  Assess the Tmax
CL/F | 168 days
  Assess the CL/F
λz | 168 days
  Assess the λz
t1/2 | 168 days
  Assess the t1/2
Vd/F | 168 days
  Assess the Vd/F
AUEC0-t of CTX-1 | 168 days
  Assess the AUEC0-t of CTX-1
Emax | 168 days
  Assess the Emax of CTX-1
TEmax | 168 days
  Assess the TEmax of CTX-1

CONTACTS AND LOCATIONS:
Overall Officials: Yanhua Ding, MD, Principal Investigator — 2nd Floor, Building 1, No. 71, Xinmin Street, Changchun, Jilin Province

IPD SHARING:
Plan to Share IPD: No